CLINICAL TRIAL: NCT02036437
Title: Titrated Oral Misoprostol Compared to Vaginal Dinoprostone for Induction of Labor: a Randomized Control Trial
Brief Title: Titrated Oral Misoprostol Compared to Vaginal Dinoprostone for Induction of Labor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sherif Essam, assistant lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: elkont1984
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Medical Induction of Labor Affecting Fetus
Keywords: Induction of Labor; Misoprostol
MeSH Terms: interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cases (Experimental): A dose of 20ug is required obtained by dissolving the 200ug tablet (Misotac® Sigma Pharmaceutical Industries) in 200 ml water (1ug per ml), the solution is shaked well before each administration. The solution will be orally administrated every two hours (max. 12 hrs) until adequate uterine contractions obtained (3 per 10 minutes each lasting 40-60 seconds) and then stopped. The initial dose will be increased to 40 ml (40ug) after two doses if there are no contractions. The timing and strength of contractions will be assessed by abdominal palpation. If the contractions are inadequate, augmentation of the active phase of labor will be attempted by hourly-titrated oral misoprostol (20 ml) +/- amniotomy.
  Interventions: Drug: Misotac® Sigma Pharmaceutical Industries
- Control (Active Comparator): Dinoprostone 3 mg (Dinoglandin® Alexandria Co. for Pharmaceuticals) will be inserted in the posterior vaginal fornix and repeated after six hours if contractions are inadequate (i.e. two doses maximum). If the contractions become inadequate, augmentation of the active phase of labor will be attempted by Syntocinon (oxytocin) infusion +/- amniotomy.
  Interventions: Drug: Dinoprostone 3 mg

INTERVENTIONS:
Drug: Misotac® Sigma Pharmaceutical Industries — The solution will be orally administrated every two hours (maximum 12 hours) until adequate uterine contractions obtained (3 per 10 minutes each lasting 40-60 seconds) and then stopped. The initial dose of 20 ml (20 ug) will be increased to 40 ml (40ug) after two doses if there are no contractions. The timing and strength of contractions will be assessed by abdominal palpation. If the contractions are inadequate, augmentation of the active phase of labor will be attempted by hourly-titrated oral misoprostol (20 ml) +/- amniotomy. If the uterine contractions are judged to be adequate, the next dose of misoprostol will be omitted.
  Other Names: Misotac (Misoprostol)
  Arms: Cases
Drug: Dinoprostone 3 mg — Dinoprostone 3 mg (Dinoglandin® Alexandria Co. for Pharmaceuticals) will be inserted in the posterior vaginal fornix and repeated after six hours if contractions are inadequate (i.e. two doses maximum). If the contractions become inadequate, augmentation of the active phase of labor will be attempted by Syntocinon (oxytocin) infusion +/- amniotomy.
  Other Names: Dinoglandin®
  Arms: Control

SUMMARY:
To test the safety and efficacy of titrated oral misoprostol compared to vaginal dinoprostone for labor induction.

DETAILED DESCRIPTION:
* There are many indications for induction of labor in the obstetric practice, of which prolonged gestational age stands as the most common indication. It is well recognized that with an unripe cervix, induction may be difficult and often unsuccessful. The use of an agent to ripen the cervix prior to induction is acceptable in the modern practice.
* Misoprostol, a prostaglandin E1 analogue, is the most interesting alternative to Dinoprostone because of its effectiveness, low cost, and temperature stability. It ripens the cervix by inducing regular uterine contractions. However, it is associated with several adverse effects especially uterine hyperstimulation, which is painful and may result in fetal compromise.
* Testing the efficacy and safety of titrated oral misoprostol versus vaginal dinoprostone may develop a new safe and effective method for labor induction.

ELIGIBILITY:
Inclusion Criteria:

* Single vertex presentation.
* Gestational age > 37 weeks calculated from last menstrual period or U/S scanning.
* Bishop score <8 .
* Not in labor.
* Reassuring fetal heart rate (CTG for 20 min on the day of induction).
* Valid indication for Induction of labor.

Exclusion Criteria:

* Gestational age <37 weeks.
* Patients with rupture of membranes.
* Previous uterine scar.
* Fetal malpresentation.
* Multiple pregnancy.
* Significant antepartum hemorrhage
* Uncontrolled DM.
* Severe Pre-eclampsia or Eclampsia
* If there are contraindications to receive the drugs, e.g. allergy, history of severe asthma,…..etc.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Induction delivery interval i.e. Time from start of medication till delivery | 24 hours

SECONDARY OUTCOMES:
Patients delivered vaginally within the first 24 hours | 24 hours
Time from start of labor augmentation by either misoprostol or Syntocinon (oxytocin) to active phase of labor | 12 hours
Duration of 1st,2nd and 3rd stages of labor | 24 hours
Maternal complications | 24 hours
  uterine hyperstimulation, postpartum hemorrhage, uterine rupture, sepsis, shivering, headache, nausea, vomiting, and retained placenta.
Mode of delivery | 24 hours
  Vaginal , instrumental or Cesarean section
Neonatal outcome | 24 hours
  Apgar score at 1 and 5 minutes and Neonatal Intensive Care Unit admission

CONTACTS AND LOCATIONS:
Overall Officials: Amr H Yehia, MD, MRCOG, Study Director — Ain Shams University
Locations (1):
- New Maternity Hospital - Ain Shams university, Cairo, Cairo Governorate, Egypt